CLINICAL TRIAL: NCT01980043
Title: Endoluminal and Needlescopic Assisted Repair of Rectal Prolapse With Abdominal Fixation Under Sedation and Local Anesthesia
Brief Title: Endoluminal and Needlescopic Assisted Repair of Rectal Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Olympus (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1209013050
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Rectal Prolapse
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rectal Prolapse (Other): endoluminal rectal prolapse repair under sedation and local anesthesia using CO2 colonoscopy to fix the rectum with sutures to the abdominal wall under needlescopic control.
  Interventions: Procedure: endoluminal rectal prolapse repair under sedation

INTERVENTIONS:
Procedure: endoluminal rectal prolapse repair under sedation — endoluminal rectal prolapse repair under sedation

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of endoluminal rectal prolapse repair under sedation and local anesthesia using CO2 colonoscopy to fix the rectum with sutures to the abdominal wall under needlescopic control. Further, investigators will evaluate the short and long-term clinical outcomes after this novel approach to treating rectal prolapse.

DETAILED DESCRIPTION:
.Aims/Objective The purpose of this study is to evaluate the safety and feasibility of endoluminal rectal prolapse repair under sedation and local anesthesia using CO2 colonoscopy to fix the rectum with sutures to the abdominal wall under needlescopic control. Further, we will evaluate the short and long-term clinical outcomes after this new procedure.

Primary Outcomes

1. Feasibility: successful completion of endoluminal rectal prolapse repair with needlescopic assistance
2. Safety: measured by the incidence of the Intraoperative complications (bowel perforation, organ injury and bleeding requiring blood transfusion)
3. Sedation and local anesthesia feasibility: surgery completed without patient intubation
4. Clinical Outcomes: rectal prolapse recurrence within 30 days, length of hospital stay and postsurgical complications
5. Long Term Clinical Outcomes: Rectal Prolapse Recurrence

Methods Design: A prospective pilot study with 10 patients who will be undergoing Combined Needlescopic and Endoluminal (Colonoscopic) Surgery under sedation and local anesthesia for Rectal Prolapse Repair with the Colon and Rectal Surgeons at WCMC. Data will be collected prospectively before, during, and after surgery.

Settings: Colon and Rectal Surgery at WCMC-NYPH Population: Patients male and female above 75 years of age, with rectal prolapse will be invited to participate in the study after surgery is deemed necessary for standard treatment of their medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age, 75 years and older, Male and Female
* BMI above 18 and ≤30
* ASA class 1-3
* willing to participate in the study

Exclusion Criteria:

* ASA class 4-5
* Previous Abdominal Surgeries including abdominal wall repair with mesh

Ages: 75 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05-20 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
rectal prolapse recurrence | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W Milsom, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical Center- NYPH, New York, New York, United States

REFERENCES:
- [Derived] Milsom JW, Trencheva K, Gadalla F, Abramovitz S, Garrett KA. Rectal Prolapse Repair with Abdominal Fixation Under Sedation and Local or Epidural Anesthesia: Prospective Pilot Study in 10 Elderly Subjects. J Laparoendosc Adv Surg Tech A. 2021 Aug;31(8):911-916. doi: 10.1089/lap.2019.0804. Epub 2020 Oct 21. PMID 33090077